CLINICAL TRIAL: NCT06033573
Title: Preoperative Assessment of Pathological Nipple Discharge With Delayed Ductal Imaging of Contrast-enhanced Spectral Mammography: an Exploratory Study
Brief Title: Preoperative Assessment of Pathological Nipple Discharge With Delayed Ductal Imaging of Contrast-enhanced Mammography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0519-01
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Nipple Discharge
Keywords: pathologic nipple discharge; contrast-enhanced spectral mammography
MeSH Terms: conditions — Galactorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contrast-enhanced spectral mammography arm (Experimental): Subjects receiving contrast-enhanced spectral mammography (CESM) 4-6 hours after the routine iopromide 370 mgI/ml-enhanced ductography
  Interventions: Diagnostic Test: contrast-enhanced spectral mammography

INTERVENTIONS:
Diagnostic Test: contrast-enhanced spectral mammography — After enrollment, subjects should undergo contrast-enhanced spectral mammography again within 4-6 hours post completing previous routine ductography to obtain a late-phase ductal image, which contains a low-energy image and a subtracted image obtained from the post processing

SUMMARY:
The goal of the prospective, interventional, self-control, open, single-center clinical study: is to evaluate the value of the delayed ductal imaging of contrast enhanced Spectral Mammography acquired in 4-6 hours after the routine iopromide 370 mgI/ml-enhanced ductography for the clinical diagnosis of patients with suspected pathologic nipple discharge.

The main questions aim to answer are:

1. Percentage of changes from baseline in imaging diagnosis caused by the results of delayed imaging.
2. The rate of reported examination-related adverse events occurred within 7 days of the delayed ductal imaging.
3. The average gland dose (AGD) of delayed ductal imaging.

After enrollment, subjects underwent CESM again within 4-6 hours post completing previous routine ductography to obtain a late-phase ductal image, which contains a low-energy image and a subtracted image obtained from the post processing.

DETAILED DESCRIPTION:
As an exploratory study, the study plans to conduct another imaging using contrast-enhanced spectral mammography (CESM) 4-6 hours after the routine iopromide 370 mgI/ml-enhanced ductography, so as to explore the optimization of the ductography technique and attempt to make a systematic description of the mammary duct structure in the Chinese population of patients with pathological nipple discharge, and thus to assess the clinical value of this delayed imaging protocol, including the effectiveness of the diagnostic dimension of the disease and the safety of the radiation dose and the degree of patient tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18-65 years old
* Completed routine iopromide 370 mgI/ml enhanced ductography for initial clinical diagnosis of suspected pathological nipple discharge, under the recommendation of the clinician
* Signed informed consent form for this study (signature and date)
* Committed to complying with study procedures and cooperating with the conducting of the full study process
* For women of childbearing age, should have taken contraceptive measures for at least one month prior to screening and must have a negative serum or urine pregnancy test, meanwhile committed to take contraceptive measures during the entire study and continue until a specified time after the end of the study

Exclusion Criteria:

* Pregnant or lactating women
* Experienced any episode of adverse events or discomfort after ductography with iopromide 370 mgI/ml
* Had any history of breast surgery, such as having undergone any invasive examination or surgical treatment due to the studied disease, including but not limited to breast duct micro-endoscopy, puncture biopsy, surgery, etc
* The ductal discharge symptom is more likely caused by other diagnosed/highly suspected diseases rather than a breast lesion, such as pituitary adenomas
* Other conditions are inappropriate for participation in this study judged by the investigator, such as the patient had difficulty to cooperate with ductography procedure, for example, loss of consciousness, communication impairment or nipple anomalies, and overly slender ducts

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of changes from baseline in imaging diagnosis caused by the results of delayed ductal imaging | 4-6 hours after the routine iopromide 370 mgI/ml-enhanced ductography
  Changes include any of the following:
  1. Changes in disease classification (based on The International Statistical Classification of Diseases, ICD-10)
  2. Any changes in the number, location and\or size (maximum and minimum diameters) of all lesions found
  3. Changes in the severity/nature of the disease with reference to the Breast Imaging Reporting and Data System classification standard

SECONDARY OUTCOMES:
Diagnostic accuracy of delayed ductal imaging results for the nature of the lesion | 4-6 hours after the routine iopromide 370 mgI/ml-enhanced ductography
  Accuracy = (Number of true positive + Number of true negative) /total number x 100% with using pathological findings as reference standard
Percentage of changes from baseline in imaging diagnosis caused by the results of delayed ductal imaging in patients with dense breasts. | 4-6 hours after the routine iopromide 370 mgI/ml-enhanced ductography
  Changes include any of the following:
  1. Changes in disease classification (based on The International Statistical Classification of Diseases, ICD-10)
  2. Any changes in the number, location and\or size (maximum and minimum diameters) of all lesions found
  3. Changes in the severity/nature of the disease with reference to the Breast Imaging Reporting and Data System classification standard
Percentage of changes from baseline in imaging diagnosis caused by the results of delayed ductal imaging in patients with non-palpable breast mass/no abnormal findings on palpation | 4-6 hours after the routine iopromide 370 mgI/ml-enhanced ductography
  Changes include any of the following:
  1. Changes in disease classification (based on The International Statistical Classification of Diseases, ICD-10)
  2. Any changes in the number, location and\or size (maximum and minimum diameters) of all lesions found
  3. Changes in the severity/nature of the disease with reference to the Breast Imaging Reporting and Data System classification standard
Kappa values for the evaluation of diagnostic imaging results of delayed ductal imaging by different radiologists. | 4-6 hours after the routine iopromide 370 mgI/ml-enhanced ductography
  Evaluate the agreement on the diagnostic evaluation of delayed images by assessors using the Kappa test.
Scores for diagnostic confidence of radiologists before and after obtaining delayed ductal imaging result. | 4-6 hours after the routine iopromide 370 mgI/ml-enhanced ductography
  on a 5-point rating scale (1-5)

OTHER OUTCOMES:
The rate of reported examination-related adverse events occurred within 7 days of delayed ductal imaging. | 7 days post delayed ductal imaging.
  Any discomfort and associated medical diagnoses post ductal imagine
The average gland dose of delayed ductal imaging. | During imaging procedure
  Total radiation of low-energy and subtracted images of delayed ductal imaging from the craniocaudal projection (CC) and the mediolateral projection (ML) of either mammary gland

CONTACTS AND LOCATIONS:
Overall Officials: Fan Yang, Dr., Principal Investigator — Union Hospital of Tongji Medical College of Huazhong University of Science and Technology
Locations (1):
- Union Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
China Policy does not allow investigator to disclose individual participant data.